CLINICAL TRIAL: NCT04637022
Title: 4K Versus 3D Laparoscopic Colporraphy by Surgeons in Training: a Prospective Randomized Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, professor, Catholic University of the Sacred Heart
Other Study IDs: DIPUSVSP-27-07-2088
Record Dates: First submitted 2020-08-31; First posted 2020-11-19 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Uterine Fibroid; Uterine Bleeding; Uterine Prolapse
Keywords: 4k laparoscopy; 3d laparoscopy; surgeons in training
MeSH Terms: conditions — Leiomyoma; Uterine Hemorrhage; Uterine Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 3D laparoscopy arm: Patients submitted to vaginal cuff closure after total laparoscopic hysterectomy using a 3D laparoscopic camera
- 4k laparoscopy arm: Patients submitted to vaginal cuff closure after total laparoscopic hysterectomy using a 4k laparoscopic camera

SUMMARY:
This prospective randomized trial aims to assess if the operative time of vaginal cuff suture performed by trainees could be reduced using 3D laparoscopy instead of 4K laparoscopy.

DETAILED DESCRIPTION:
All patients with benign uterine pathology at preoperative examinations (pelvic ultrasound and / or magnetic resonance and / or CT) and with indication for total laparoscopic hysterectomy with consequently need for laparoscopic suture of the vaginal cuff, will be enrolled in the study.

- I TIME/OUT OF PROTOCOL TIME (performed by expert surgeons) While under general anesthesia, the patient is positioned in the dorsal lithotomic position with both legs supported in stirrups with a Trendelenburg tilt and arms along the body. A four disposable or reusable, sterile trocar transperitoneal approach is used. A 10 mm port is inserted at the umbilicus for the telescope. Once pneumoperitoneum (12 mmHg) is achieved, intra-abdominal visualization will be obtained with a 0° 4K high-definition telescope (VISERA UHD 4K 10 mm, Olympus Winter & IBE GMBH, Hamburg - Germany) or with 0° 3D laparoscopy high-definition (Olympus Winter & IBE GMBH, Hamburg - Germany).

Two additional 5 mm ports are placed under direct visualization, in the right lower abdomen medial to the right obliterated umbilical artery and in the left lower abdomen lateral to the inferior epigastric vessels. One more 5-mm trocar is inserted in the right mid abdomen at the level of the umbilicus. The instruments used include bipolar grasper, monopolar scissors, monopolar hook, various graspers and a suction irrigation system. Clermont Ferrand uterine manipulator (Model K.Storz Endoskope,Tuttlingen, Germany) is optionally used to move the uterus.

Total hysterectomy is then performed according to standard technique.

- II TIME/PROTOCOL TIME (performed by surgeon in training) The vaginal vault is closed with a 0 Vycril suture laparoscopically (continuous suture). In order to avoid excess operating time, 15 min was allocated for completion of cuff closure by surgeons-in-training, after which time the attending surgeon took over this task.

Operative time, estimated blood loss, incidence of intra or post-operative complications, postoperative pain, days of hospitalization and costs will be recordered

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from benign gynecological pathology (uterine fibromatosis, abnormal blood loss, complex hyperplasia with atypia, uterine prolapse) with indication for total uterine hysterectomy and consequently need for laparoscopic suture of the vaginal cuff
* American Society of Anesthesiologists (ASA) class < 3
* Patient's informed consent

Exclusion Criteria:

* Suspected neoplastic pathology
* Patients not eligible for surgery
* Actual pregnancies or pelvic inflammatory disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with benign uterine pathology at preoperative examinations (pelvic ultrasound and / or magnetic resonance and / or CT) and with indication for total laparoscopic hysterectomy with consequently need for laparoscopic suture of the vaginal cuff, will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-09-10 (Estimated); Study Completion 2021-09-10 (Estimated)

PRIMARY OUTCOMES:
operative time | intra-operative
  To compare the time taken to close the vaginal cuff, which was defined as time, starting from the initial grasp of the suture to cutting the suture, with 3D Laparoscopy vs 4K laparoscopy

SECONDARY OUTCOMES:
Intra-operative complications | intra-operative
  Evaluate the incidence of intraoperative complications in the two laparoscopic system (intraoperative blood loss, need for intraoperative transfusions, bladder lesions, ureteral lesions, vascular lesions, intestinal lesions)

OTHER OUTCOMES:
post-operative complications | up to 3 months
  - Evaluate the incidence of postoperative complications (dehiscence of the vaginal cuff, fever, urinary tract infections, surgical wound infections)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli, IRCCS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided